CLINICAL TRIAL: NCT03789279
Title: RATATOUILLE Study (inteRnATional hAnd funcTiOn stUdy Following dIstaL radiaL accEss)
Brief Title: Observational Study of Hand Function After Distal Transradial Access for Angiography
Acronym: RATATOUILLE
Status: Completed | Type: Observational
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: MC Zuiderzee (Unknown)
Responsible Party: Principal Investigator, Dr Thomas J Ford, Honorary Clinical Lecturer, University of Glasgow
Other Study IDs: 18-WS-0182; 245250 (Other: IRAS)
Record Dates: First submitted 2018-12-26; First posted 2018-12-28 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Radial Artery Occlusion; Nerve Injury
Keywords: Invasive coronary angiography; Distal transradial arterial access; Anatomical snuffbox; dTRA; dRA; Distal radial; Radial artery occlusion
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Distal transradial arterial access: Patients undergoing invasive coronary angiography via the distal radial approach (anatomical snuffbox)

SUMMARY:
Traditionally, coronary angiograms are performed through the radial artery which is accessed above the palm of the 'right' hand. In recent years, some cardiologists are performing this procedure from the back of the wrist in as the radial artery courses through the anatomical snuffbox (distal radial access). The aim of this study is to determine the prevalence of hand dysfunction following coronary angiography via the distal radial artery.

DETAILED DESCRIPTION:
In this multi centre observational registry, we will recruit patients undergoing planned invasive coronary angiography. Inclusion criteria include:

1. Age ≥ 18 years.
2. The distal radial artery must be palpable and non-occlusive flow must be confirmed by Doppler ultrasound.
3. Patient should be able to comply with the protocol.
4. Provide written informed consent before study participation.

The primary endpoint is the overall prevalence of hand dysfunction defined as any significant reduction from baseline score in any of the following five domains:

DASH score Levine Katz score VAS score Sensory function Pinch grip strength.

Specifically hand function will be assessed at 4 time points using simple tests of hand strength, sensation and ultrasound to assess the arterial latency.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. The distal radial artery must be palpable and non-occlusive flow must be confirmed by Doppler ultrasound.
3. Patient should be able to comply with the protocol.
4. Provide written informed consent before study participation.

Exclusion Criteria:

1. Obligatory femoral or forearm radial access
2. Previous ipsilateral forearm radial artery occlusion.
3. Undergoing another procedure involving the ipsilateral radial artery, performed between the index procedure and the follow-up date.
4. Enrolment in another study that competes or interferes with this study.
5. Poor clinical condition like cardiogenic shock, that prohibits pre- and postprocedural function tests.
6. Any other condition which, in the opinion of the investigator or operator, may pose a significant hazard to the subject if he or she is enrolled in the study.
7. Co-morbidity that excludes patient follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients for inclusion are those by whom coronary angiography or angioplasty is indicated as part of clinical decision-making or therapy. Operators with adequate experience at the discretion of the principal investigator in distal radial access are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of hand dysfunction | 1 month
  Any significant deterioration from baseline in hand function according to the 5 studied domains.

SECONDARY OUTCOMES:
Success of distal radial access | Day 0
  Successful introduction of sheath
Vascular access complications (other than occlusion and bleeding) | Day 0
  Surgical complications or clinically important vascular access complications
Puncture time | Day 0
  Time from skin puncture to successful placement of wire into the artery
Radial artery occlusion - including level of occlusion (prox/distal) | 0-12 months
  USS guide
Fluoroscopy time | Day 0
  Minutes
Hemostasis duration | Day 0
  Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Kiemeneij, MD, Principal Investigator — MC Zuiderzee; Ahmed Hassan, MD, Study Director — MC Zuiderzee
Locations (1):
- University of Glasgow/Golden Jubilee Research Foundation, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No